CLINICAL TRIAL: NCT02185300
Title: A Phase 1, Single Dose, Crossover, Relative Bioavailability Study of a Dolutegravir Dispersible Tablet as Compared to a Dolutegravir Pediatric Granule Formulation and Effect of Different Types of Water on the Dispersible Tablet in Healthy Volunteers(200401)
Brief Title: Bioavailability Study of a Dolutegravir Dispersible Tablet and Effect of Different Types of Water on the Dispersible Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 200401
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-09

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK1349572; granule; pediatric; CONTREX mineral water; free-acid; chelating; cations; divalent; dolutegravir; dispersible tablet; relative bioavailability
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sequence ABCDE (Experimental): Subject will be administered treatments in the sequence ABCDE where, A = Single dose of DTG 20 mg of the pediatric granule formulation reconstituted with purified water; B = Single dose of DTG 20 mg DT dispersed in LMC water; C = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water; D= Single dose of DTG 20 mg DT dispersed in LMC water, held for 30 minutes(mins), re-dispersed, and then taken by subject; E = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water, held for 30 minutes, re-dispersed, and then taken by subject
  Interventions: Drug: Dolutegravir Pediatric Granules; Drug: Dolutegravir Dispersible Tablet
- Sequence BCDEA (Experimental): Subject will be administered treatments in the sequence BCDEA where, A = Single dose of DTG 20 mg of the pediatric granule formulation reconstituted with purified water; B = Single dose of DTG 20 mg DT dispersed in LMC water; C = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water; D= Single dose of DTG 20 mg DT dispersed in LMC water, held for 30 mins, re-dispersed, and then taken by subject; E = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water, held for 30 mins, re-dispersed, and then taken by subject
  Interventions: Drug: Dolutegravir Pediatric Granules; Drug: Dolutegravir Dispersible Tablet
- Sequence CDEAB (Experimental): Subject will be administered treatments in the sequence CDEAB where, A = Single dose of DTG 20 mg of the pediatric granule formulation reconstituted with purified water; B = Single dose of DTG 20 mg DT dispersed in LMC water; C = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water; D= Single dose of DTG 20 mg DT dispersed in LMC water, held for 30 mins, re-dispersed, and then taken by subject; E = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water, held for 30 mins, re-dispersed, and then taken by subject
  Interventions: Drug: Dolutegravir Pediatric Granules; Drug: Dolutegravir Dispersible Tablet
- Sequence DEABC (Experimental): Subject will be administered treatments in the sequence DEABC where, A = Single dose of DTG 20 mg of the pediatric granule formulation reconstituted with purified water; B = Single dose of DTG 20 mg DT dispersed in LMC water; C = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water; D= Single dose of DTG 20 mg DT dispersed in LMC water, held for 30 mins, re-dispersed, and then taken by subject; E = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water, held for 30 mins, re-dispersed, and then taken by subject
  Interventions: Drug: Dolutegravir Pediatric Granules; Drug: Dolutegravir Dispersible Tablet
- Sequence EABCD (Experimental): Subject will be administered treatments in the sequence EABCD where, A = Single dose of DTG 20 mg of the pediatric granule formulation reconstituted with purified water; B = Single dose of DTG 20 mg DT dispersed in LMC water; C = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water; D= Single dose of DTG 20 mg DT dispersed in LMC water, held for 30 mins, re-dispersed, and then taken by subject; E = Single dose of DTG 20 mg DT dispersed in CONTREX mineral water, held for 30 mins, re-dispersed, and then taken by subject
  Interventions: Drug: Dolutegravir Pediatric Granules; Drug: Dolutegravir Dispersible Tablet

INTERVENTIONS:
Drug: Dolutegravir Pediatric Granules — Dolutegravir pediatric granules are supplied as 40 grams bulk bottles containing 0.4% weight by weight of dolutegravir to be reconstituted with 73 mL of purified water to yield a dolutegravir concentration of 1.6 milligram / millilitre. 12.5 mL of reconstituted granules contain 20 mg DTG
Drug: Dolutegravir Dispersible Tablet — Dolutegravir is available as 5mg dispersible tablets and can be administered as 4 tablets dispersed in 12.5 mL LMC water and consumed immediately or 4 tablets dispersed in 12.5 mL CONTREX mineral water and consumed immediately or 4 tablets dispersed in 12.5 mL LMC water, allow to stand at room temperature for 30 mins, re-suspend mixture and consumed or 4 tablets dispersed in 12.5 mL CONTREX mineral water, allow to stand at room temperature for 30 mins, re-suspend mixture and consumed

SUMMARY:
Dolutegravir (DTG) is an HIV-1 integrase inhibitor approved in the United States, Canada, Australia and EU. A dispersible tablet has been developed for pediatric use as an alternative to the granule formulation, already in development, and the approved film-coated tablet. This is a single-center, randomized, open-label, 5-way crossover study in healthy adult subjects. The study will evaluate the relative bioavailability of five dosing regimens: 20 mg DTG pediatric granules (Treatment A) and of DTG 20 mg dispersible tablets (DTG 20 mg DT) after dispersed in: low mineral content(LMC) water (Treatment B); dispersed in CONTREX™ mineral water (Treatment C); dispersed in low mineral content water and consumed after standing for 30 minutes (Treatment D) and dispersed in CONTREX mineral water and consumed after standing for 30 minutes (Treatment E). Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug. CONTREX is a trademark of Nestlé Waters Corporation.

ELIGIBILITY:
Inclusion Criteria

* Males or females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agree and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight +/- 50 kilogram (kg) for males and +/- 45 kg for females and body mass index (BMI) within the range 18.5 - 31.0 kilogram/square meter (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, bilateral salpingectomy, bilateral oophorectomy or hysterectomy for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter (mIU/mL) and estradiol < 40 picograms per milliliter (pg/ml) (<147 picomole/liter [pmol/L]) is confirmatory. Child-bearing potential with negative pregnancy test as determined by serum or urine human chorionic gonadotropin (hCG) test at screening and prior to dosing AND agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 5 days post-last dose OR have only same-sex partners, when this is her preferred and usual lifestyle.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine transaminase (ALT), alkaline phosphatase and bilirubin <= 1.5x upper limit of the normal range (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat from screening to period 1, day -1 is allowed for eligibility determination.
* QT duration corrected for heart rate (QTc) < 450 millisecond (msec), using Bazett Correction Formula, QT correction using Bazett Formula (QTcB). A single repeat from screening to period 1, day -1 is allowed for eligibility determination.

Exclusion Criteria:

* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Lactating females.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Regular use of tobacco- or nicotine-containing products within 60 days prior to screening.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject's systolic blood pressure is outside the range of 90-140 millimeters of mercury (mmHg), or diastolic pressure is outside the range of 45-90 mmHg, or heart rate is outside the range of 50-100 beats per minute (bpm) for female subjects or 45-110 bpm for male subjects. A single repeat from screening to period 1, day -1 is allowed for eligibility determination.
* Exclusion criteria for screening electrocardiogram (ECG) (a single repeat is allowed for eligibility determination): Heart rate - For males <45 and >110 bpm and for females <50 and >100 bpm, PR Interval <120 and >220 msec, QRS duration <70 and >120 msec, QTc interval (Bazett) >450 msec, evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization), any clinically significant arrhythmia which, in the opinion of the investigator and GSK Medical Monitor, will interfere with the safety for the individual subject, or any conduction abnormality with the exception of 1st degree atrioventricular block or incomplete right bundle branch block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters following single dose administration of DTG 20 mg DT dispersed in LMC water | Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose), Day 2 (24 hours) and Day 3 (48 hours)
  PK parameters include area under the concentration-time curve from time zero extrapolated to infinite time (AUC [0-infinity]) Maximum observed concentration (Cmax) and apparent oral clearance (CL/F)
Composite of PK parameters following single dose administration of DTG 20 mg DT dispersed in CONTREX mineral water | Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose), Day 2 (24 hours) and Day 3 (48 hours)
  PK parameters include AUC (0-infinity), Cmax and CL/F
Composite of PK parameters following single dose administration of DTG 20 mg DT dispersed in LMC water with 30-minute holding | Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose), Day 2 (24 hours) and Day 3 (48 hours)
  PK parameters include AUC (0-infinity), Cmax and CL/F

SECONDARY OUTCOMES:
Composite of PK parameters following single dose administration of DTG 20 mg DT dispersed in LMC water | Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose), Day 2 (24 hours) and Day 3 (48 hours)
  PK parameters include area under the plasma concentration-time curve from time of dose administration to time of last quantifiable post-dose sample [AUC(0-t)]; observed concentration at 24h post-dose (C24); terminal elimination phase half-life (t½); lag time for absorption (tlag); and time to maximum observed concentration (tmax)
Composite of PK parameters following single dose administration of DTG 20 mg DT dispersed in CONTREX mineral water | Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose), Day 2 (24 hours) and Day 3 (48 hours)
  PK parameters include AUC(0-t), C24; t½; tlag; and tmax will be evaluated for DTG 20 mg DT
Composite of PK parameters following single dose administration of DTG 20 mg DT dispersed in LMC water with 30-minute holding | Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose), Day 2 (24 hours) and Day 3 (48 hours)
  PK parameters include AUC(0-t), C24; t½; tlag; and tmax
Composite of PK parameters following single dose administration of DTG 20 mg DT in CONTREX mineral water with 30-minute holding | Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose), Day 2 (24 hours) and Day 3 (48 hours)
  PK parameters include AUC (0-infinity), Cmax, CL/F, AUC(0-t); C24; t½; tlag; and tmax
Palatability of DTG 20 mg DT | Day 1 (Period 1 only)
  Palatability questionnaire containing 11 questions will be administered to each subject within 10 minutes following the dose of DTG (Period 1 only)
Safety as assessed by number of subjects with adverse events, change from baseline in vital signs and as toxicity grading of clinical laboratory tests | Up to 14 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Vital signs include blood pressure and heart rate. Clinical laboratory parameters will include hematology and clinical chemistry

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States